CLINICAL TRIAL: NCT02559583
Title: Hemato-Oncology Latin America Observational Registry in CLL, Multiple Myeloma, Non-Hodgkin Lymphoma
Brief Title: Observational Study in Participants With Chronic Lymphocytic Leukemia (CLL), Multiple Myeloma (MM) and Non-Hodgkin's Lymphoma (NHL) in Latin America
Acronym: HOLA
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR105066; PCI-32765MMY4001 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2015-04-23; First posted 2015-09-24 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Multiple Myeloma; Leukemia; Lymphoid; Lymphoma; Non-Hodgkin
Keywords: Multiple Myeloma; chronic lymphocytic leukemia; Non-Hodgkin lymphoma
MeSH Terms: conditions — Multiple Myeloma; Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — non-Hodgkin's lymphoma protocol 8503

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Participants with Chronic Lymphocytic Leukemia (CLL): This is an observational study. Data will be captured for Participant's with diagnosis of Chronic Lymphocytic Leukemia according to hospital records in the questionnaire provided by the Sponsor.
  Interventions: Other: Chronic Lymphocytic Leukemia (CLL)
- Participants with Multiple Myeloma (MM): This is an observational study. Data will be captured for Participant's with diagnosis of Multiple Myeloma (MM) according to hospital records in the questionnaire provided by the Sponsor.
  Interventions: Other: Multiple Myeloma (MM)
- Participants with Non-Hodgkin's lymphoma (NHL): This is an observational study. Data will be captured for Participant's with diagnosis of non-Hodgkin's lymphoma (NHL) data according to hospital records in the questionnaire provided by the Sponsor.
  Interventions: Other: Non-Hodgkin's lymphoma (NHL)

INTERVENTIONS:
Other: Chronic Lymphocytic Leukemia (CLL) — This is observational study. Participants with Chronic Lymphocytic Leukemia (CLL) will be observed for 1 year.
  Groups: Participants with Chronic Lymphocytic Leukemia (CLL)
Other: Multiple Myeloma (MM) — This is observational study. Participants with Multiple Myeloma (MM) will be observed for 1 year.
  Groups: Participants with Multiple Myeloma (MM)
Other: Non-Hodgkin's lymphoma (NHL) — This is observational study. Participants with non-Hodgkin's lymphoma (NHL) will be observed for 1 year.
  Groups: Participants with Non-Hodgkin's lymphoma (NHL)

SUMMARY:
The primary purpose of the study is to quantify participants' demographic parameters, country standard therapies, treatment patterns and outcomes among participants with chronic lymphocytic leukemia (CLL), multiple myeloma (MM) and non-Hodgkin's lymphoma (NHL) in oncology concentration hospitals in Latin America.

DETAILED DESCRIPTION:
This is a retrospective (take a look back at events that already have taken place), non-interventional, multicenter (when more than one hospital or medical school team work on a medical research study) study to review medical records of adult participants with a diagnosis of CLL, MM or NHL anytime since 01 January 2006. Only data available from clinical practice will be collected. All eligible participants at participating centers will be included regardless of participant's demographics, prior or current treatments for disease, or clinical outcome. The period of observation will span from 01 January 2006 through present, but all eligible participants must be followed for a minimum of 1 year, unless the participant died within that first year. Participant demographic parameters, standard therapies, treatment patterns and outcomes will be primarily quantified.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic lymphocytic leukemia (CLL), multiple myeloma (MM), or non-Hodgkin lymphoma (NHL) anytime since January 1, 2006
* At least one year of data following first observed diagnosis except in the case of the participant death within one year following first observed diagnosis
* Participant must sign a participation agreement/informed consent form (ICF)

Exclusion Criteria:

- Having one and only one consult in the center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic lymphocytic leukemia (CLL), multiple myeloma (MM) and non-Hodgkin's lymphoma (NHL) in oncology concentration hospitals in Latin America
Sampling Method: Probability Sample
Enrollment: 5443 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Previous Comorbidities | 1 year
  Comorbidities included: heart, diabetes, hypertension, renal, infections, other neoplasia, neurologic, rheumatologic, HIV, thrombosis, bone and other.
Number of Participants as per treatment therapy received | 1 year
  Cancer treatment (Chronic Lymphocytic Leukemia [CLL], Multiple Myeloma [MM] and non-Hodgkin lymphoma [NHL]) for all participants is summarized by the number of participants who had any type of surgery or radiotherapy (external radiation or brachytherapy) or other drug treatments.
Overall survival | 1 year
  Overall Survival (OS) was defined as the time from date of starting treatment to death due to any cause.
Number of Participants with Response to Treatment | 1 year
  Number of participants who responded to treatment is presented. Treatment response will be assessed based on complete response or partial response.

SECONDARY OUTCOMES:
Incidence Percentage of Participants with Chronic Lymphocytic Leukemia (CLL), Multiple Myeloma (MM) and non-Hodgkin lymphoma (NHL) | 1 year
  Incidence of CLL, MM and NHL will be reported. It is a percentage of the population at risk of developing the disease.
Prevalence Percentage of Participants with CLL, MM and NHL | 1 year
  Prevalence of CLL, MM and NHL will be reported. Prevalence will be estimated using available population demographic information as the denominators and using the percentage of registered participants with those cancers at the sites as the numerators.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (23):
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - La Plata Lpl Lpl
- Brazil (6):
  - Belo Horizonte
  - Fortaleza
  - Goiânia
  - Porto Alegre
  - São José do Rio Preto
  - São Paulo
- Santiago, Chile
- Colombia (5):
  - Bogotá
  - Bogotá Dc
  - Cali
  - Floridablanca
  - Medellín
- Guatemala City, Guatemala
- Mexico (5):
  - Huixquilucan
  - Mexico City
  - México
  - Monterrey
  - Toluca
- Panama (2):
  - Panama City
  - Panama Republic Panama

REFERENCES:
- [Derived] Chiattone C, Gomez-Almaguer D, Pavlovsky C, Tuna-Aguilar EJ, Basquiera AL, Palmer L, de Farias DLC, da Silva Araujo SS, Galvez-Cardenas KM, Gomez Diaz A, Lin JH, Chen YW, Machnicki G, Mahler M, Parisi L, Barreyro P. Real-world analysis of treatment patterns and clinical outcomes in patients with newly diagnosed chronic lymphocytic leukemia from seven Latin American countries. Hematology. 2020 Dec;25(1):366-371. doi: 10.1080/16078454.2020.1833504. PMID 33095117